CLINICAL TRIAL: NCT06992492
Title: Vojta Reflex Versus Lung Squeezing Technique In Preterm Neonate With Respiratory Distress Syndrome
Brief Title: Vojta Reflex Versus Lung Squeezing Technique in Respiratory Distress Preterm Neonate
Acronym: RDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman mustafa mohammed elsagheer, Physiotherapist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FPTBSUREC/0905/2325
Record Dates: First submitted 2025-05-05; First posted 2025-05-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Distress Syndrome
Keywords: RDS; preterm neonates
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): Group A infants will receive reflex rolling technique along with conventional chest physical therapy (postural drainage, percussion and vibration) plus medical treatment with special emphasis on whether Surfactant therapy is given or not. This maneuver includes a slight rotation of the head towards the side from which the stimulus is delivered. The starting position for performing the first phase of reflex rolling is the asymmetric supine position, with the limbs freely lying on the resting surface. A digit pressure will exert on the chest area, where the mammillary line crosses the insertion of the diaphragm, either at the level of the 6th rib, or between the 5th and the 6th, or between the 6th and the 7th. Each treatment consists in delivering four stimuli, two to the left half of the chest (stimulations I and II) and two to the right half of the chest (stimulations III and IV). Each stimulus will be consisted of slight pressure, progressively oriented in dorsal, medial and crani
  Interventions: Procedure: vojta therapy +conventional chest physical therapy
- group B (Active Comparator): Group B infants will receive lung squeezing technique along with conventional chest physiotherapy (postural drainage, percussion and vibration) plus medical treatment with special emphasis on whether Surfactant therapy is given or not. Lung squeeze technique consists of 3- cumulative chest compressions lasting for 5 seconds, followed by a gentle low "release phase", with the chest wall completely released; the second compressions are performed successively for5 minutes on one hemithorax, then 5 minutes on the other hemi thorax. The infant will be in supine position, and without body tilt, for a total of 10 minutes. Use both hands to perform the squeeze on one hemithorax at one time. Place One hand on the posterolateral aspect of the hemi thorax and the other hand covered the anterior chest extending from the lower ribs to above the clavicle of the infant
  Interventions: Procedure: lung squeezing technique +conventional chest physical therapy
- group C (Active Comparator): Conventional Chest Physical Therapy will be given for both the groups A and B and for group C in isolation manner with medical treatment with special emphasis on whether Surfactant therapy is given or not.it includes postural drainage, vibration, and percussion. Postural drainage will be applied to infants by elevating head of the infant at 30 degrees to prevent gastro esophageal reflex and aspiration. In neonates and infants 'tenting' (using the first three or four fingers of one hand with slight elevation of the middle finger). Chest percussion will be given with motion from the wrist. Vibration of the chest will be done manually by placing the fingers on the chest wall over the segment being drained and the wrist and the elbow remained immobile, isometrically contracting the muscles of the forearm and hand to cause a vibratory motion. The procedure will be performed for 5min. Chest percussion position lying down on the right side and on the left, with 5 min duration on each sid
  Interventions: Procedure: conventional chest physical therapy

INTERVENTIONS:
Procedure: vojta therapy +conventional chest physical therapy — infants will receive reflex rolling technique along with conventional chest physical therapy (postural drainage, percussion and vibration) plus medical treatment with special emphasis on whether Surfactant therapy is given or not. This maneuver includes a slight rotation of the head towards the side from which the stimulus is delivered. The starting position for performing the first phase of reflex rolling is the asymmetric supine position, with the limbs freely lying on the resting surface. A digit pressure will exert on the chest area, where the mammillary line crosses the insertion of the diaphragm, either at the level of the 6th rib, or between the 5th and the 6th, or between the 6th and the 7th. Each treatment consists in delivering four stimuli, two to the left half of the chest (stimulations I and II) and two to the right half of the chest (stimulations III and IV). Each stimulus will be consisted of slight pressure, progressively oriented in dorsal, medial and cranial direct
  Arms: group A
Procedure: lung squeezing technique +conventional chest physical therapy — infants will receive lung squeezing technique along with conventional chest physiotherapy (postural drainage, percussion and vibration) plus medical treatment with special emphasis on whether Surfactant therapy is given or not. Lung squeeze technique consists of 3- cumulative chest compressions lasting for 5 seconds, followed by a gentle low "release phase", with the chest wall completely released; the second compressions are performed successively for5 minutes on one hemithorax, then 5 minutes on the other hemi thorax. The infant will be in supine position, and without body tilt, for a total of 10 minutes. Use both hands to perform the squeeze on one hemithorax at one time. Place One hand on the posterolateral aspect of the hemi thorax and the other hand covered the anterior chest extending from the lower ribs to above the clavicle of the infant.
  Arms: group B
Procedure: conventional chest physical therapy — Conventional Chest Physical Therapy will be given for both the groups A and B and for group C in isolation manner with medical treatment with special emphasis on whether Surfactant therapy is given or not.it includes postural drainage, vibration, and percussion. Postural drainage will be applied to infants by elevating head of the infant at 30 degrees to prevent gastro esophageal reflex and aspiration. In neonates and infants 'tenting' (using the first three or four fingers of one hand with slight elevation of the middle finger). Chest percussion will be given with motion from the wrist. Vibration of the chest will be done manually by placing the fingers on the chest wall over the segment being drained and the wrist and the elbow remained immobile, isometrically contracting the muscles of the forearm and hand to cause a vibratory motion. The procedure will be performed for 5min. Chest percussion position lying down on the right side and on the left, with 5 min duration on each side
  Arms: group C

SUMMARY:
The goal of this clinical trial study is to find out the difference in the effect of vojta therapy and lung squeezing technique on preterm neonate with respiratory distress syndrome, to investigate the effect of vojta therapy and lung squeezing technique on Oxygen saturation and Respiratory rate, to evaluate the effect of vojta therapy and lung squeezing technique on (The length of hospital stay, Silverman Anderson score, Downe's score for respiratory distress syndrome (RDS) in preterm neonate. The main question it aims to answer is:

Is There a significant difference in the effect of vojta therapy and lung squeezing technique in preterm neonate with respiratory distress syndrome. Researchers will compare effect of vojta therapy and lung squeezing technique and control group. neonates diagnosed with respiratory distress syndrome aged from 28 to 36 weeks will be recruited for this study for three weeks from neonate intensive care unit.

neonates will receive conventional chest physical therapy for the control group and convetional chest physical therapy plus vojta therapy or lung squeezing technique for the two other groups twice daily for three weeks.

DETAILED DESCRIPTION:
Type of study: randomized clinical trial. this study is a prospective interventional study one that will be conducted on 90 preterm neonates of both sexes from Neonatal Intensive care unit in Beni-Suef university, their gestational age ranged from 28 to 36 weeks and randomly divided into 3 equal groups:

1. study group (A) include preterm neonates with respiratory distress syndrome will receive vojta therapy along with conventional chest physical therapy (postural drainage, percussion and vibration) plus medical treatment with special emphasis on whether Surfactant therapy is given or not.
2. study group (B) include preterm neonates with respiratory distress syndrome will receive lung squeezing technique along with conventional chest physical therapy (postural drainage, percussion and vibration) plus medical treatment with special emphasis on whether Surfactant therapy is given or not.
3. control group (C) include preterm neonates with respiratory distress syndrome will receive conventional chest physical therapy (postural drainage, percussion and vibration) plus medical treatment only with special emphasis on whether Surfactant therapy is given or not.

Measurement procedures:

1.) Oxygen saturation and Respiratory rate: For the three study groups, the SpO2 and respiratory rate will be measured and noted before the reflex stimulation, at the end of stimulation II, at the end of stimulation IV and at 5, 15, 25 minutes after the whole series of stimulations, during each of the twice daily treatments. Throughout the whole procedure, the NBs were continuously monitored with a Vismo PVM-2701 monitor to assess any adverse effect, including hypoxemia (SpO2 < 90) which would indicate suspension of the technique. physiotherapist followed the infants for three weeks.

Study variables: 1)RR = assessed by clinical evaluation of chest movement in one minute and SpO2 = measured with a pulse oximeter.

2) Silverman Anderson score: The Silverman Andersen Respiratory Severity Score (RSS) evaluates five parameters of work of breathing and assigns an overall score with a patient breathing comfortably a "0" and a patient in severe respiratory distress a "10".

Score 0-3 = Mild respiratory distress - O2 by hood Score 4-6 = Moderate respiratory distress - CPAP Score > 6 = Impending respiratory failure

3) Downe's score for RDS: Downe score is an objective method to assess the severity of respiratory distress in newborns. It includes respiratory rate (RR), recessions, grunt, air entry and fractional oxygen requirement. Each parameter is score on a scale of 0, 1 and 2 with increasing severity. Total score ranges from 0 to 10.Score:

* <4 = follow up.
* 4-7 = clinical respiratory distress; monitor arterial blood gases.
* 7 = respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates will be:

  * Ranging from 28-36 weeks of gestation admitted to NICU with diagnosis of respiratory distress syndrome (RDS)on oxygen therapy.
  * Medically free from any other diseases except RDS.
  * On CPAP for respiratory support.

Exclusion Criteria:

* Preterm neonates who meet one of the following criteria will be excluded:

  * Musculoskeletal disorders
  * Encephalopathy
  * Recent surgery
  * Neonates with respiratory and cardiac congenital anomalies
  * mechanically ventilated
  * genetic syndromes
  * segmental or lobar collapse confirmed on chest X-ray
  * congenital malformation
  * asphyxia at birth
  * treatment with neurotrophic drugs
  * intraventricular hemorrhage < 2 grade

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | from enrollment for three weeks twice daily
  Oxygen saturation (SpO2) will be measured and noted before the reflex stimulation, at the end of stimulation II, at the end of stimulation IV and at 5, 15, 25 minutes after the whole series of stimulations, twice daily. Throughout the whole procedure, oxygen saturation will be continuously monitored with a Vismo PVM-2701 monitor to assess any adverse effect, including hypoxemia (SpO2 < 90), which would indicate suspension of the technique. physiotherapist will follow the infants for three weeks.
respiratory rate | from enrollment for three weeks twice daily
  respiratory rate will be measured and noted before the reflex stimulation, at the end of stimulation II, at the end of stimulation IV and at 5, 15, 25 minutes after the whole series of stimulations, twice daily. Throughout the whole procedure, the respiratory rate will be continuously monitored with a Vismo PVM-2701 monitor to assess any adverse effect which would indicate suspension of the technique. physiotherapist will follow the infants for three weeks.

SECONDARY OUTCOMES:
Silverman Anderson score | at the start of the study and after the intervention once day for three weeks
  The Silverman Andersen Respiratory Severity Score (RSS) evaluates five parameters of work of breathing and assigns an overall score with a patient breathing comfortably a "0" and a patient in severe respiratory distress a "10".
  Score 0-3 = Mild respiratory distress - O2 by hood Score 4-6 = Moderate respiratory distress - CPAP Score > 6 = Impending respiratory failure
Downe's score for RDS | at the start of the study and after the intervention once day for three weeks
  Downe score is an objective method to assess the severity of respiratory distress in newborns. It includes respiratory rate (RR), recessions, grunt, air entry and fractional oxygen requirement. Each parameter is score on a scale of 0, 1 and 2 with increasing severity. Total score ranges from 0 to 10.
  Score:
  * <4 = follow up.
  * 4-7 = clinical respiratory distress; monitor arterial blood gases.
  * 7 = respiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Sherine H Mehani, professor, Study Director — Beni-Suef University
Locations (2):
- Egypt (2):
  - Beni-Suef university hospitals, Banī Suwayf
  - Beni_Suef university, Banī Suwayf

IPD SHARING:
Plan to Share IPD: No